CLINICAL TRIAL: NCT03611478
Title: Examining the Effects of One-Month Probiotic Treatment on Mental Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Principal Investigator, Andrew Scholey, Professor, Swinburne University of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NH-03884
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Mental Fatigue; Cognitive Function; Mood
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Half the participants will receive the probiotic formulation while the other half will receive placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind trial, with randomisation being conducted by a disinterested third party. Unblinding will not occur until data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic formulation (Experimental): Contains a probiotic formulation. One capsule to be taken by mouth once daily for 28 days.
  Interventions: Dietary Supplement: Probiotic formulation
- Placebo (Placebo Comparator): Matching placebo to be taken once daily by mouth for 28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic formulation — Probiotic capsule
  Arms: Probiotic formulation
Dietary Supplement: Placebo — Placebo capsule identical in taste and appearance to probiotic capsule
  Arms: Placebo

SUMMARY:
The aim of this study is to demonstrate the effects of 28-days supplementation with a novel probiotic formulation on mental fatigue following a cognitive load in healthy adults. Half of the participants will receive the probiotic formulation while the other half will receive placebo.

DETAILED DESCRIPTION:
A total of 128 participants will be recruited to take part in this trial.

The supplement contains selected strains of lactobacilli and bifidobacteria which have been well studied in human clinical trials. Previous clinical trials have demonstrated improvements in cognitive function and mood after supplementation with various combinations of lactobacilli and bifidobacteria.

The specific strains present in the current investigation have been studied in a number of clinical trials in which no adverse events were linked to the strains. The benefits of probiotic supplements on health is well established, and has led to an increase in use, as well as the addition of probiotic strains in dietary supplements. Despite this, only a small number of controlled trials have directly investigated the cognitive benefits associated with probiotic supplementation.

The current study therefore aims to investigate the anti-fatigue effects of a probiotic supplement after a period of cognitive demand. We will be measuring the effects of the probiotic supplement compared to a placebo using assessments of mental fatigue, cognition, memory and mood.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-50 years, inclusive.
2. Willing and able to provide written informed consent.
3. Ability of the participant (in the Principal Investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
4. Agreement to comply with the protocol and study restrictions.
5. Available for all study visits.
6. Females of child-bearing potential required to provide a negative urine pregnancy test and be using effective contraception (e.g. surgically sterilized (tubal ligation or hysterectomy or partner is post-vasectomy, with sterility confirmed) or use an IUD (intrauterine device), a diaphragm or condom combined with contraceptive sponge, foam or jelly, or be using an oral contraceptive (the pill) for at least 2 cycles before the Screening-visit (Visit 0)).
7. Fluent in written and spoken English.
8. In good general health as judged by the Investigator/Clinical advisor based on medical history.
9. Must have normal, or corrected to normal vision.
10. Body mass index between 18.5 and 29.9kg/m2 (inclusive).
11. Participant is willing to maintain habitual diet (including caffeine and alcohol) and physical activity patterns throughout the study period.
12. Participant is willing and able to comfortably abstain from caffeine for 10 hours prior to and throughout the test visits, (2-3 hours).
13. Participant is willing to abstain from alcohol for 12 hours and vigorous physical activity for 12 hours prior to all study visits.

Exclusion Criteria:

1. History of dementia, stroke and other neurological conditions.
2. Traumatic loss of consciousness in the last 12 months.
3. History of epilepsy or Parkinson's disease.
4. Formal diagnosis of anxiety, depression or any psychiatric disorder that the Principal Investigator believes would interfere with the objectives of the study and requiring treatment (prescription of antidepressant, antipsychotic or other long term medication and/or referral for long term psychotherapy) in the last 2 years. Brief interventions for normal life events such as exam anxiety or bereavement are not an exclusion.
5. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal (irritable bowel syndrome (IBS), inflammatory bowel disease (IBD)), immunological, metabolic (including diabetes or cardiovascular disease), endocrine or bleeding disorders, neurodevelopmental or any condition which contraindicates, in the Principal Investigator's judgement, entry to the study.
6. Uncontrolled hypertension (systolic blood pressure > 160mm Hg or diastolic blood pressure >100 mm Hg).
7. Currently taking (from day of screening onwards) or have previously taken (last 4 weeks prior to screening) psychoactive medication (anxiolytics, sedatives, hypnotics, anti-psychotics, anti-depressants, anti-convulsants, centrally acting corticosteroids, opioid pain relievers).
8. Currently taking (from day of screening onwards) medication that the Principal Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results such as:

   * high dose anticoagulant medication such as warfarin, heparin, clopidogrel, dabigatran, ticagrelor
   * non-steroidal anti-inflammatory drugs (NSAIDS; excluded only for daily use)
   * over-the-counter sleep medication (not categorized as sedatives, hypnotics or anti-depressants)
   * anti-cholinergic drugs or acetylcholinesterase inhibitors: bethanechol (Urecholine), donepezil (Aricept), rivastigmine (Exelon), galantamine (Reminyl), neostigmine (Prostigmin)
   * anti-histamines that cause drowsiness (eg. Ranitidine)
   * pseudoephedrine and phenylephrine
9. Currently taking (from day of screening onwards) dietary supplements that the Principal Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results such as: melatonin, vitamin E, multivitamins, B vitamin complex, ginkgo biloba, fish oil, St. John's Wort or other cognitive enhancing dietary or herbal supplements over the study period.
10. Recent (within last 4 weeks prior to screening) or ongoing antibiotic therapy during the intervention period.
11. Daily consumption of concentrated sources of probiotics and/or prebiotics within 2 weeks of screening and throughout the intervention period other than the provided study products (e.g., probiotic/prebiotic tablets, capsules, drops or powders or yoghurts/yoghurt drinks containing probiotics).
12. Pregnant or lactating female, or pregnancy planned during intervention period.
13. Have self-reported dyslexia.
14. Current misuse of alcohol, drugs, or prescription medication.
15. Current smoker.
16. Self-declared illicit drug users (including cannabis and cocaine) for 3 weeks prior to screening and during the intervention period.
17. Excessive alcohol consumption (drinking on 5 or more days a week) for 3 weeks prior to screening and during the intervention period.
18. Contraindication to any substance in the investigational product.
19. Participation in another study with any investigational product within 30 days of screening and during the intervention period.
20. Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study.
21. Participant under administrative or legal supervision.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Mental fatigue score (VAS-mental fatigue) | 28 days
  Difference in mental fatigue score as the participant moves through six cycles of a cognitive demand battery (CDB). The cognitive demand battery consists of three tasks (RVIP, serial threes and serial sevens, described below), and is designed to increase cognitive load. Six cycles of the battery are completed in succession at each testing visit. The mental fatigue scale (VAS-mental fatigue) is completed after each cycle of the CDB (6 times over the course of one hour, per visit). Participants rate their level of mental fatigue on a 100-mm scale from "not at all" to "extremely". The primary outcome is difference in mental fatigue score (VAS-mental fatigue) as the participant moves through the six cycles of the CDB, (after cognitive load) absolute change from baseline (Visit 2) to 28 days (Visit 3) between the active vs placebo group.

SECONDARY OUTCOMES:
RVIP number correct | 28 days
  Percentage of target strings correctly detected on the rapid visual information processing (RVIP) task throughout each of the six cycles of the CDB. In this task, which lasts for 5 minutes, a series of numbers rapidly appear on the screen one at a time. Participants are instructed to press the space bar whenever they detect a sequence of either 3 consecutive odd or 3 consecutive even numbers.
RVIP reaction time | 28 days
  Average reaction time for correct detections (RVIP) throughout each of the six cycles of the CDB.
RVIP false alarms | 28 days
  The number of false alarms (RVIP) throughout each of the six cycles of the CDB
Serial threes subtraction total | 28 days
  Total number of subtractions on the serial threes subtraction task, regardless of whether correct or incorrect, throughout each of the six cycles of the CDB. In this two minute task, participants are given a starting number and instructed to subtract three from this number. They must then type in the number they are left with and press enter. After this no numbers are visible but the participant must continue to subtract three and enter their responses.
Serial threes errors | 28 days
  Total number of incorrect subtractions (serial threes subtraction task) throughout each of the six cycles of the CDB
Serial sevens total | 28 days
  Total number of subtractions (serial sevens subtraction task) throughout each of the six cycles of the CDB. This task is the same as the serial threes task, except that participants must subtract seven instead of three.
Serial sevens errors | 28 days
  Total number of errors (serial sevens subtraction task) throughout each of the six cycles of the CDB
Immediate word recall - correct | 28 days
  The number of correctly identified words in the immediate word recall task. Participants see a list of 15 words that they are instructed to remember. After seeing the last word, the participant has 60 seconds to write down as many of the words as they can remember.
Immediate word recall - errors | 28 days
  The number of errors in the immediate word recall task (words not included in the original list)
Immediate word recall - intrusions | 28 days
  The number of intrusions in the immediate word recall task (words similar to those included in the original list but not identical).
Delayed word recall - Correct | 28 days
  The number of correctly identified words in the delayed word recall task. After completing the CDB (approximately one hour after presentation of the 15 words), the participant has 60 seconds to write down as many of the words as they can remember from the original list.
Delayed word recall - errors | 28 days
  The number of errors in the delayed word recall task (words not included in the original list)
Delayed word recall - intrusions | 28 days
  The number of intrusions in the delayed word recall task (words similar to those included in the original list but not identical).
Delayed word recognition - reaction time | 28 days
  Mean reaction time to word recognition in delayed word recognition task following cognitive load. After participants have viewed the word list and completed the immediate word recall task, they complete the CDB which lasts for one hour. On completion of the CDB, participants complete a word recognition task. In this task, the original 15 target words plus an additional 15 distractor words are presented one at a time, in a randomized order. Participants are instructed to indicate whether or not they recognize the word from the original list by pressing the 'Yes' or 'No' button as appropriate as quickly as possible, mean reaction times are measured in msec.
Word recognition - original words accuracy | 28 days
  Accuracy of responses (%) to original target words in delayed word recognition task following cognitive load (CDB).
Word recognition - distractor words accuracy | 28 days
  Accuracy of responses (%) to novel distractor words in delayed word recognition following cognitive load (CDB).
Self-reported alertness score | 28 days
  Participants are presented with a number of 100-mm visual analogue scales (Bond-Lader mood scales) where they indicate their current feelings. The alertness score is calculated by averaging scores on lines anchored by alert-drowsy, attentive-dreamy, lethargic-energetic, muzzy-clearheaded, well-coordinated-clumsy, mentally slow-quick witted, strong-feeble, interested-bored, incompetent-proficient. This is completed before and after the CDB.
Self-reported contentment score | 28 days
  Participants are presented with a number of 100-mm visual analogue scales (Bond-Lader mood scales) where they indicate their current feelings. The contentment score is calculated by averaging scores on lines anchored by contented-discontented, troubled-tranquil, happy-sad, antagonistic-friendly, withdrawn-sociable. This is completed before and after the CDB.
Self-reported calmness score | 28 days
  Participants are presented with a number of 100-mm visual analogue scales (Bond-Lader mood scales) where they indicate their current feelings. The calmness score is calculated by averaging scores on lines anchored by calm-excited, tense-relaxed. This is completed before and after the CDB.
Difference in self-reported stress score (VAS-stress) before and after a cognitive load | 28 days
  The Stress Visual Analogue Scale (VAS-Stress) consists of a single 100 mm line with end-points labelled 'Not at all' and 'Very much so'. Participants are instructed to mark the line, depending on how "stressed" they feel at that point in time. This is completed twice in each session, once prior to the CDB, and once after the battery is complete. The difference between pre- and post-CDB score is calculated, and the difference is compared between baseline and 28 days.
Self-reported stress score (VAS-stress) - pre-CDB only | 28 days
  The Stress Visual Analogue Scale (VAS-Stress) consists of a single 100 mm line with end-points labelled 'Not at all' and 'Very much so'. Participants are instructed to mark the line, depending on how "stressed" they feel at that point in time. The pre-CDB score is compared between baseline and 28 days to provide an assessment of stress without cognitive load.
Difference in self-reported physical fatigue score (VAS-fatigue) before and after a cognitive load | 28 days
  The Physical Fatigue Visual Analogue Scale (VAS-fatigue) consists of a single 100 mm line with end-points labelled 'Not at all' and 'Very much so'. Participants are instructed to mark the line, depending on how "physically fatigued" they feel at that point in time. This is completed twice in each session, once prior to the CDB, and once after the battery is complete. The difference between pre- and post-CDB score is calculated, and the difference is compared between baseline and 28 days.
Self-reported physical fatigue score (VAS-fatigue) - pre-CDB only | 28 days
  The Physical Fatigue Visual Analogue Scale (VAS-Fatigue) consists of a 100 mm line with end-points labelled 'Not at all' and 'Very much so'. Participants are instructed to mark the line, depending on how "physically fatigued" they feel at that point in time. The pre-CDB score is compared between baseline and 28 days to provide an assessment of physical fatigue without cognitive load.
Self-reported state anxiety (STAI) before and after a cognitive load | 28 days
  The 'State' subscale of the STAI contains 20 items, and requires participants to rate how much they feel like each item at the time of response. The scale is scored on a 4-point scale ranging from 'not at all' to 'very much so'. Scores range from 20 to 80, with higher scores indicating higher levels of anxiety. Participants will be required to complete the state version of the STAI twice per session, once before the commencement of the CDB, and once at completion.
Mental fatigue score on the Chalder Fatigue Scale | 28 days
  The 14-item Chalder Fatigue Scale (CFS) measures both physical and mental fatigue, as well as a total fatigue rating, on a 4-point scale ranging from 'better than usual' to 'much worse than usual'.
Physical fatigue score on the Chalder Fatigue Scale | 28 days
  The 14-item CFS measures both physical and mental fatigue, as well as a total fatigue rating, on a 4-point scale ranging from 'better than usual' to 'much worse than usual'.
Total fatigue score on the Chalder Fatigue Scale | 28 days
  The 14-item CFS measures both physical and mental fatigue, as well as a total fatigue rating, on a 4-point scale ranging from 'better than usual' to 'much worse than usual'.
Self-reported sleep quality - total score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported duration of sleep score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported sleep disturbance score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported sleep latency score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported daytime dysfunction score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported habitual sleep efficiency score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Subjective sleep quality score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported use of sleep medications score | 28 days
  The Pittsburgh Sleep Quality Index (PSQI) was originally designed to measure sleep quality and disturbance in clinical populations, and has been subsequently utilized in a number of research settings. The PSQI is a self-rated scale measured over a one-month interval. The scale is comprised of 19 individual items that generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction. The scale also has five items to be answered by a bed partner, if applicable, but these answers are not included in the scoring of the scale. For the current study, these five questions will be removed from the scale.
Self-reported vitality score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported physical functioning score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported bodily pain score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported general health perceptions score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported physical role functioning score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported emotional role functioning score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported social role functioning score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported mental health score (SF-36) | 28 days
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. The SF-36 will be completed once per session.
Self-reported depression score (DASS-21) | 28 days
  The Depression, Anxiety and Stress scale (DASS-21) is a 21-item questionnaire that is split into three factors: depression, anxiety and stress. The DASS-21 is made up of affect-related questions pertaining to both physical (e.g. 'dry mouth') and mood symptoms (e.g. 'down-hearted'). Each item is scored on a 4-point scale from 0 to 3, with higher scores indicating a higher degree of dysfunction. It is important to note that lower scores reflect a lack of symptoms and not a more positive mood. Furthermore, as the experience of such symptoms is common in every-day life, the DASS-21 is considered suitable for use in non-clinical settings.
Self-reported anxiety score (DASS-21) | 28 days
  The Depression, Anxiety and Stress scale (DASS-21) is a 21-item questionnaire that is split into three factors: depression, anxiety and stress. The DASS-21 is made up of affect-related questions pertaining to both physical (e.g. 'dry mouth') and mood symptoms (e.g. 'down-hearted'). Each item is scored on a 4-point scale from 0 to 3, with higher scores indicating a higher degree of dysfunction. It is important to note that lower scores reflect a lack of symptoms and not a more positive mood. Furthermore, as the experience of such symptoms is common in every-day life, the DASS-21 is considered suitable for use in non-clinical settings.
Self-reported stress score (DASS-21) | 28 days
  The Depression, Anxiety and Stress scale (DASS-21) is a 21-item questionnaire that is split into three factors: depression, anxiety and stress. The DASS-21 is made up of affect-related questions pertaining to both physical (e.g. 'dry mouth') and mood symptoms (e.g. 'down-hearted'). Each item is scored on a 4-point scale from 0 to 3, with higher scores indicating a higher degree of dysfunction. It is important to note that lower scores reflect a lack of symptoms and not a more positive mood. Furthermore, as the experience of such symptoms is common in every-day life, the DASS-21 is considered suitable for use in non-clinical settings.
Self-reported confrontive coping score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported distancing score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported self-controlling score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported seeking social support score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported accepting responsibility score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported escape-avoidance score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported planful problem-solving score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Self-reported positive re-appraisal score (WAYS) | 28 days
  The Ways of Coping Questionnaire (WAYS) is a 66-item scale designed to measure an individual's ability to cope with stress over the past week. The scale measures coping processes, not coping styles. The scale is divided into 8 subscales; confrontive coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, planful problem solving, positive re-appraisal. The scale is completed once per session.
Positive effects of on-trial experiences | 28 days
  At the completion of the trial, participants will be asked an open-ended question about any positive effects they may have experienced on their physical or mental health during the study, to allow qualitative analysis of on-trial experiences.
Negative effects of on-trial experiences | 28 days
  At the completion of the trial, participants will be asked an open-ended question about any negative effects they may have experienced on their physical or mental health during the study, to allow qualitative analysis of on-trial experiences.
Unusual effects of on-trial experiences | 28 days
  At the completion of the trial, participants will be asked an open-ended question about any unusual effects they may have experienced on their physical or mental health during the study, to allow qualitative analysis of on-trial experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Scholey, PhD, Principal Investigator — Swinburne University of Technology
Locations (1):
- Centre for Human Psychopharmacology, Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No